CLINICAL TRIAL: NCT06837961
Title: The Effects of Lactococcus Lactis JCM 5805 (LC-Plasma) Lactic Acid Bacteria on Immune Response and Reducing Symptoms of Upper Respiratory Infectious Disease in Australian Healthy Adults. Randomized Placebo-controlled Double-blind Parallel Group Study.
Brief Title: LC-Plasma on Immune Response and Reducing Symptoms of Upper Respiratory Infectious Diseases
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: RDC Clinical Pty Ltd (Industry)
Collaborators: Kirin Holdings Company, Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GU/2025/073
Record Dates: First submitted 2025-02-17; First posted 2025-02-20 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-02

CONDITIONS: Healthy Volunteer; Immune Response
Keywords: LC-Plasma; Healthy volunteer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LC-Plasma (Experimental): 1 tablet containing 50mg LC-Plasma is taken daily for 4 weeks
  Interventions: Dietary Supplement: LC-Plasma
- Placebo (Placebo Comparator): 1 tablet containing 50mg microcrystalline cellulose is taken daily for 4 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: LC-Plasma — 1 tablet containing 50mg LC-Plasma is taken daily for 4 weeks
  Arms: LC-Plasma
Other: Placebo — 1 tablet containing 50mg MCC is taken daily for 4 weeks
  Arms: Placebo

SUMMARY:
The goal of this study is to evaluate the effects of LC-Plasma on the innate and acquired immune systems, including the activation of pDCs, which play a role in virus elimination, as well as to assess its efficacy in reducing clinical symptoms of upper respiratory infectious diseases in healthy adults. Researchers will compare LC-Plasma to placebo, participants will take a tablet containing LC-Plasma or placebo daily for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who can provide a signed and dated informed consent form after confirming their willingness to participate.
* Individuals willing to comply with all study procedures during the study period, including daily monitoring record compliance, cooperating with blood and urine sample collection and performing regular RATs.
* Healthy people living in Australia aged 18-60 (both men and women).
* Individuals who have received at least two doses of a SARS-CoV-2 vaccine, with at least two weeks having passed since the last dose.
* Individuals who are not currently infected with SARS-CoV-2 and, if previously infected, have recovered and have been infection-free for at least four weeks.
* Individuals who do not have any chronic or acute illnesses, including respiratory and/or gastrointestinal and/or other diseases, (e.g. hypertension, IBS, IBD, SLE, cancer, asthma, primary or secondary immunodeficiencies etc.), at the time of enrolment.

Exclusion Criteria:

* Individuals medically prescribed medications that would affect the immune and/or the inflammatory response.
* Individuals deemed unsuitable for participation by Griffith CTU staff and/or the study clinician.
* Active smokers/vapers and/or individuals with nicotine or drug habits.
* Individuals currently participating in (or planning to participate in) other clinical trials.
* Women who are pregnant, planning to become pregnant during the study period, or are currently breastfeeding.
* Individuals unable to abstain from alcohol for two days prior to blood and urine sample collection.
* Individuals unable to refrain from consuming other lactic acid bacteria supplements.
* Individuals who are known to be HIV, HTLV-1, or HCV positive (based on answers to the enrolment questionnaire).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 241 (Actual)
Dates: Start 2025-04-29 (Actual); Primary Completion 2025-11-03 (Actual); Study Completion 2025-11-03 (Actual)

PRIMARY OUTCOMES:
The degree of activation of plasmacytoid dendritic cells (pDCs) | Week 0 to week 4
  The degree of activation of plasmacytoid dendritic cells (pDCs) is measured using the indicators CD304+/CD123+, CD86+, or HLA-DR+

SECONDARY OUTCOMES:
Activation of Cytotoxic T Lymphocytes (CTLs) | Week 0 to week 4
  The evaluation of CTLs responsible for virus elimination will be determined using the indicator (CD8+/CD3+/CD4-/IFN-γ+).
Anti-viral Activity of PBMCs | Week 0 to week 4
  The anti-viral activity gene expression and IFN-α & β production capability of PBMCs, both unstimulated and mildly stimulated with CpG, will be measured.
WURSS-24 Symptom Score | Week 0 to week 4
  Symptoms will be measured using the Wisconsin Upper Respiratory Symptom Survey (WURSS-24)
Rapid antigen test (RAT) | Week 0 to week 4
  Rapid antigen test (RAT) for Flu A/B, RSV & SARS-CoV-2. Will be conducted by participants once per week, with additional tests if symptoms are present.

OTHER OUTCOMES:
Safety: Occurrence of adverse events | Week 0 to week 4
  Occurrence of adverse events
Safety: Confirmation of medical history during study period | Week 0 to week 4
  Confirmation of medical history during study period

CONTACTS AND LOCATIONS:
Overall Officials: Yusuke Ushida, Study Director — Kirin Holdings Company, Limited; Osamu Kanauchi, Study Director — Kirin Holdings Company, Limited
Locations (1):
- Griffith University, Southport, Queensland, Australia

IPD SHARING:
Plan to Share IPD: Undecided